CLINICAL TRIAL: NCT04410016
Title: Evaluation of a Workplace Intervention to Implement Supported COVID-19 Wellbeing Centres in a Healthcare Workplace During and After the Coronavirus Pandemic: The COVID-WELL Study
Brief Title: Evaluation of Staff COVID-19 Wellbeing Centres in a Healthcare Workplace: COVID-WELL Study
Acronym: COVID-WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Holly Blake, Dr Holly Blake, Associate Professor of Behavioural Science, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COVID-WELL_May20
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: All staff have access to the Staff Wellbeing Centres (usual practice). In this study the investigators will conduct a questionnaire survey with all Nottingham University Hospitals National Health Service (NHS) staff about their mental wellbeing, and use of this facility. The investigators will conduct qualitative interviews with users and non-users of the Wellbeing Centres (staff) as well as the Wellbeing Buddies (support workers).
Masking Description: This is an evaluation of a service - the Wellbeing Centres at Nottingham University Hospitals National Health Service (NHS) Trust - which are a form of 'intervention' for staff provided during the coronavirus pandemic. Therefore the investigators will conduct interviews with people who have used the centres, or who have acted as support workers within them. The investigators will survey all staff in the Trust, and interview up to 45 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staff Wellbeing Centre (Experimental): Wellbeing Centres are rooms where staff employed at the hospital trust can go for a break, rest, relaxation, quiet time out, advice support or signposting. They are manned by Wellbeing Buddies who are support workers who offer advice and signposting services. The Centres are accessible to all staff at the Trust.
  Interventions: Other: Staff Wellbeing Centres

INTERVENTIONS:
Other: Staff Wellbeing Centres — 2 Centres (rooms) accessible to staff for rest and relaxation, work breaks, supports advice and signposting. They are manned by support workers called Wellbeing Buddies.

SUMMARY:
Evaluation of a workplace intervention to implement supported wellbeing centres in a healthcare workplace during and after the COVID-19 pandemic.

Mixed-Methods Evaluation study - including collection of service use monitoring data, online survey and qualitative interviews.

DETAILED DESCRIPTION:
Project Aims:

1. To describe the cost, reach and usage of the Staff Wellbeing Centres
2. To gather insight into experiences of those who access the facility ('service users') as well as those of support workers ('wellbeing buddies').
3. To identify any facilitators, obstacles or barriers to accessing the facility.
4. To identify perceptions of facility users and non-users towards the value of the facilities during and after the coronavirus pandemic.
5. To establish recommendations for longer-term sustainability of the wellbeing centres.

Interviews will be conducted with up to 45 interview participants (10-15 Wellbeing Buddies, 25-30 Staff).

Online survey will be conducted - all Nottingham University Hospitals National Health Service (NHS) staff invited to take part (>14,000).

The survey will include measures of mental wellbeing (Warwick-Edinburgh Wellbeing Scale, 14-item - license received), and single items measures of job stressfulness, job satisfaction, presenteeism, turnover intentions and work engagement.

ELIGIBILITY:
Inclusion Criteria:

* National Health Service staff which includes employees, volunteers or healthcare students, as well as bank staff (all have access to the Staff Wellbeing Centres).
* Ability to give informed consent. For survey element: Ability to access the internet (to complete the online survey) For interview element: Ability to attend an individual interview.

Exclusion Criteria:

• Inability to communicate in spoken English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale | Baseline
  14-item scale to measure mental wellbeing. Total scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.

SECONDARY OUTCOMES:
Single Item Measure of Global Job Stressfulness (Houdmont et al, 2019) | Baseline
  Single-item measure. Scores range from 1 to 5 and higher scores indicated greater job stressfulness.
Single Item Global Job Satisfaction Measure (Dolbier et al, 2005) | Baseline
  Single-item measure. Scores range from 1 to 5 and higher scores indicated greater job satisfaction.
Single Item Measure of Presenteeism (Aronsson & Gustafsson, 2004) | Baseline
  Single-item measure. Scores range from 1 to 4, with higher scores indicating greater presenteeism.
Single Item Measure of Turnover intentions (Ryan et al, 2017) | Baseline
  Single-item measure. Scored 1=no intent to leave, 2=intent to leave
Work Engagement (Shaufeli et al, 2006) | Baseline
  Dedication subscale of the 9-item Utrecht Work Engagement Scale (3 items will be used: 2, 3 and 4). Scores range from 0 to 6, with higher scores indicating greater work engagement.

OTHER OUTCOMES:
Qualitative Interviews with Staff | Once per study, telephone interview (during a 6-week interview period)
  Users and non-users of Wellbeing Centres
Qualitative Interviews with Wellbeing Buddies | Once per study, telephone interview (during a 6-week interview period)
  Support Workers within the Wellbeing Centres

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Interview data will be made available on request (after study end).
Time Frame: Interview data will be available on request at study end (after publication of findings).
Access Criteria: On request.

REFERENCES:
- [Result] Blake H, Gupta A, Javed M, Wood B, Knowles S, Coyne E, Cooper J. COVID-Well Study: Qualitative Evaluation of Supported Wellbeing Centres and Psychological First Aid for Healthcare Workers during the COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Mar 31;18(7):3626. doi: 10.3390/ijerph18073626. PMID 33807306
- [Result] Blake H, Yildirim M, Wood B, Knowles S, Mancini H, Coyne E, Cooper J. COVID-Well: Evaluation of the Implementation of Supported Wellbeing Centres for Hospital Employees during the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Dec 15;17(24):9401. doi: 10.3390/ijerph17249401. PMID 33333913
- See also: departmental news item — https://www.nottingham.ac.uk/healthsciences/news/the-covid-well-study.aspx